CLINICAL TRIAL: NCT00422422
Title: Open-Label, Single-Arm, Multicenter, Pharmacokinetic, Safety, and Efficacy Study of Adjunctive Administration of Brivaracetam in Subjects From ≥1 Month to <16 Years Old With Epilepsy
Brief Title: Open-label, Pharmacokinetic, Safety and Efficacy Study of Adjunctive Brivaracetam in Children With Epilepsy.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N01263; 2006-006536-22 (EudraCT Number)
Expanded Access: NCT03532516 (Available)
Record Dates: First submitted 2007-01-10; First posted 2007-01-17 (Estimated); Results first posted 2017-01-09 (Estimated); Last update posted 2018-07-11 (Actual); Status verified 2016-11

CONDITIONS: Epilepsy
Keywords: Brivaracetam; Epilepsy; Child; Pharmacokinetics; Adolescents
MeSH Terms: conditions — Epilepsy | interventions — brivaracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Brivaracetam (Experimental)
  Interventions: Drug: Brivaracetam

INTERVENTIONS:
Drug: Brivaracetam — Oral solution
  Evaluation period (3 weeks up-titration):
  For subjects ≥8 years:
  * ~0.4 mg/kg bid for Week 1
  * ~0.8 mg/kg bid for Week 2
  * ~1.6 mg/kg bid for Week 3
  For subjects <8 years:
  * ~0.5 mg/kg bid for Week 1
  * ~1.0 mg/kg bid for Week 2
  * ~2.0 mg/kg bid for Week 3
  Down-titration period (up to 2 weeks):
  For subjects ≥8 years:
  * ~0.8 mg/kg bid for Week 4
  * ~0.4 mg/kg bid for Week 5
  For subjects <8 years:
  * ~1.0 mg/kg bid for Week 4
  * ~0.5 mg/kg bid for Week 5

SUMMARY:
Initial study in children with epilepsy to evaluate the pharmacokinetics, safety, tolerability and preliminary efficacy of adjunctive treatment with brivaracetam, and to develop dosing adaptations for future studies.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of epilepsy
* Subject having at least 1 seizure (any type) during the 3 weeks before first visit
* Stable dosing of 1-3 concomitant antiepileptic drugs

Exclusion Criteria:

* Pregnant or nursing females
* Concomitant use of Levetiracetam
* Epilepsy secondary to a Progressive cerebral disease/tumor or other neurodegenerative disease
* History of status epilepticus
* Clinically significant acute or chronic illness, underlying disease or medication condition
* History of suicide attempt

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2011-07; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (39):
- United States (12):
  - 108, Gulf Breeze, Florida
  - 110, Miami, Florida
  - 103, Wellington, Florida
  - 106, Boston, Massachusetts
  - 101, Saint Paul, Minnesota
  - 113, Chesterfield, Missouri
  - 105, Buffalo, New York
  - 104, Rochester, New York
  - 107, Cincinnati, Ohio
  - 114, Pittsburgh, Pennsylvania
  - 109, Nashville, Tennessee
  - 117, Houston, Texas
- Belgium (3):
  - 202, Brussels
  - 203, Brussels
  - 201, Leuven
- Czechia (3):
  - 502, Hradec Králové
  - 504, Ostrava Porubo
  - 501, Prague
- Mexico (7):
  - 602, Aguascalientes
  - 611, Chihuahua City
  - 609, Ciuliacan
  - 603, Guadalajara
  - 604, Mexico City
  - 610, Monterrey
  - 607, San Luis Potosí City
- Poland (8):
  - 404, Bialystok
  - 403, Gdansk
  - 406, Kielce
  - 402, Krakow
  - 401, Poznan
  - 408, Rzeszów
  - 407, Szczecin
  - 405, Wroclaw
- Spain (6):
  - 309, Barcelona
  - 306, Madrid
  - 301, Palma de Mallorca
  - 304, Santander
  - 308, Valencia
  - 303, Zaragoza

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The N01263 study began recruitment in July 2011, with subjects enrolled in the European Union, Mexico, and the United States. The study concluded in March 2013.
Groups:
- Brivaracetam (ES): Brivaracetam (BRV) was given as 2 equally divided oral doses twice daily (bid). The dosage was adjusted as following:
  For subjects ≥8 years:
  * 0.4 mg/kg bid for Week 1
  * 0.8 mg/kg bid for Week 2
  * 1.6 mg/kg bid for Week 3
  For subjects <8 years:
  * 0.5 mg/kg bid for Week 1
  * 1.0 mg/kg bid for Week 2
  * 2.0 mg/kg bid for Week 3
  Down-titration period (up to 2 weeks):
  For subjects ≥8 years:
  * 0.8 mg/kg bid for Week 4
  * 0.4 mg/kg bid for Week 5
  For subjects <8 years:
  * 1.0 mg/kg bid for Week 4
  * 0.5 mg/kg bid for Week 5
Period: Overall Study
Arm/Group | Brivaracetam (ES)
Started | 100
Completed | 90
Not Completed | 10
Not completed — Lack of Efficacy | 1
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 2
Not completed — SAE, non-fatal | 1
Not completed — AE, non-serious non-fatal | 5

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics consists of the Enrolled Subjects analysis set, which is comprised of all subjects enrolled into the study.
Arm/Group | Brivaracetam (ES)
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.3 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 49
Weight [Mean (Standard Deviation); unit: kilograms] | 24.2 (16.2)
Height [Mean (Standard Deviation); unit: centimeters] | 111.8 (32.9)
BMI [Median (Standard Deviation); unit: kg/m^2] | 17.1 (3.4)
Racial Group [Number; unit: participants]
  Black or African American | 4
  White | 80
  Other | 16

OUTCOME MEASURES:

1. Primary Outcome: Mean Trough Plasma Concentration at 3rd Level for Age Range ≥1 Month to <2 Years
Time Frame: Day 21
Measure: Mean (Standard Deviation); unit: ug/mL
Groups:
- Brivaracetam (PPS): Brivaracetam (BRV) was given as 2 equally divided oral doses twice daily (bid). The dosage was adjusted as following:
  For subjects ≥8 years:
  * 0.4 mg/kg bid for Week 1
  * 0.8 mg/kg bid for Week 2
  * 1.6 mg/kg bid for Week 3
  For subjects <8 years:
  * 0.5 mg/kg bid for Week 1
  * 1.0 mg/kg bid for Week 2
  * 2.0 mg/kg bid for Week 3
  Down-titration period (up to 2 weeks):
  For subjects ≥8 years:
  * 0.8 mg/kg bid for Week 4
  * 0.4 mg/kg bid for Week 5
  For subjects <8 years:
  * 1.0 mg/kg bid for Week 4
  * 0.5 mg/kg bid for Week 5
Arm/Group | Brivaracetam (PPS)
Number analyzed (Participants) | 12
ug/mL | 0.825 (0.826)

2. Primary Outcome: Mean Trough Plasma Concentration at 3rd Level for Age Range ≥2 to <12 Years
Time Frame: Day 21
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Brivaracetam (PPS)
Number analyzed (Participants) | 22
ug/mL | 0.967 (0.536)

3. Primary Outcome: Mean Trough Plasma Concentration at 3rd Level for Age Range ≥12 to <16 Years
Time Frame: Day 21
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Brivaracetam (PPS)
Number analyzed (Participants) | 4
ug/mL | 1.117 (0.400)

4. Primary Outcome: Mean Max Plasma Concentration for Age Range ≥1 Month to <2 Years
Time Frame: Day 21
Measure: Mean (Full Range); unit: ug/mL
Arm/Group | Brivaracetam (PPS)
Number analyzed (Participants) | 12
ug/mL | 2.071 [0.320 to 4.305]

5. Primary Outcome: Mean Max Plasma Concentration for Age Range ≥2 to <12 Years
Time Frame: Day 21
Measure: Mean (Full Range); unit: ug/mL
Arm/Group | Brivaracetam (PPS)
Number analyzed (Participants) | 22
ug/mL | 2.673 [0.561 to 5.418]

6. Primary Outcome: Mean Max Plasma Concentration for Age Range ≥12 to <16 Years
Time Frame: Day 21
Measure: Mean (Full Range); unit: ug/mL
Arm/Group | Brivaracetam (PPS)
Number analyzed (Participants) | 4
ug/mL | 2.861 [2.627 to 3.371]

7. Secondary Outcome: Number of Subjects With at Least One Treatment-emergent Adverse Event Reported During the 3-week Evaluation Period
Time Frame: Baseline to end of the 3-week evaluation period
Measure: Number; unit: participants
Groups:
- Brivaracetam (SS): Brivaracetam (BRV) was given as 2 equally divided oral doses twice daily (bid). The dosage was adjusted as following:
  For subjects ≥8 years:
  * 0.4 mg/kg bid for Week 1
  * 0.8 mg/kg bid for Week 2
  * 1.6 mg/kg bid for Week 3
  For subjects <8 years:
  * 0.5 mg/kg bid for Week 1
  * 1.0 mg/kg bid for Week 2
  * 2.0 mg/kg bid for Week 3
  Down-titration period (up to 2 weeks):
  For subjects ≥8 years:
  * 0.8 mg/kg bid for Week 4
  * 0.4 mg/kg bid for Week 5
  For subjects <8 years:
  * 1.0 mg/kg bid for Week 4
  * 0.5 mg/kg bid for Week 5
Arm/Group | Brivaracetam (SS)
Number analyzed (Participants) | 99
participants | 66

8. Secondary Outcome: Number of Subjects With a 50 % Reduction in Seizures Based on Seizure Diary Data From Baseline to End of the 3-week Evaluation Period
Time Frame: Baseline to end of the 3-week evaluation period
Measure: Number; unit: participants
Groups:
- Brivaracetam (FAS): Brivaracetam (BRV) was given as 2 equally divided oral doses twice daily (bid). The dosage was adjusted as following:
  For subjects ≥8 years:
  * 0.4 mg/kg bid for Week 1
  * 0.8 mg/kg bid for Week 2
  * 1.6 mg/kg bid for Week 3
  For subjects <8 years:
  * 0.5 mg/kg bid for Week 1
  * 1.0 mg/kg bid for Week 2
  * 2.0 mg/kg bid for Week 3
  Down-titration period (up to 2 weeks):
  For subjects ≥8 years:
  * 0.8 mg/kg bid for Week 4
  * 0.4 mg/kg bid for Week 5
  For subjects <8 years:
  * 1.0 mg/kg bid for Week 4
  * 0.5 mg/kg bid for Week 5
Arm/Group | Brivaracetam (FAS)
Number analyzed (Participants) | 80
participants | 17

9. Secondary Outcome: Percent Compliance With Brivaracetam Oral Solution During the 3-week Evaluation Period
Time Frame: Baseline to the end of the 3-week evaluation period
Population: Although 99 subjects were in the Safety Set and confirmed to have taken at least one dose of BRV, details on study drug intake were not able to be collected for 2 subjects. Therefore compliance could only be calculated for 97 subjects.
Measure: Number; unit: participants
Arm/Group | Brivaracetam (SS)
Number analyzed (Participants) | 97
participants
  <80 % | 5
  80 % to 120 % | 90
  >120 % | 2

ADVERSE EVENTS:
Time Frame: Treatment-emergent Adverse Events (TEAEs) were collected during the course of the study up to day 49.
Description: The Safety Set is all enrolled subjects who took at least 1 dose of study drug.
  Subjects had the ability to report more than one event. The Serious Adverse Events and Non-serious Adverse Events sections are reported in this manner.
Arm/Group | Brivaracetam (SS)
Serious Adverse Events (participants affected / at risk) | 8/99
Other Adverse Events (participants affected / at risk) | 33/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brivaracetam (SS) (N=99)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1)
Toxoplasmosis (Infections and infestations) | 1 (1)
Cytomegalovirus test positive (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Convulsion (Nervous system disorders) | 4 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brivaracetam (SS) (N=99)
Irritability (General disorders) | 8 (9)
Pyrexia (General disorders) | 7 (8)
Fatigue (General disorders) | 5 (5)
Pharyngotonsillitis (Infections and infestations) | 5 (5)
Decreased appetite (Metabolism and nutrition disorders) | 7 (7)
Somnolence (Nervous system disorders) | 8 (9)
Convulsion (Nervous system disorders) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 but <= 180 days to review results communications prior to public release and may delete information that is confidential and compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that the results shall be published regardless of outcome.